CLINICAL TRIAL: NCT00041639
Title: A Phase I/II Study of Radioimmunotherapy With 90Y-Humanized MN-14 IgG Administered as a Single Dose to Patients With Refractory Advanced/Metastatic Pancreatic Carcinoma
Brief Title: Safety Study of 90Y-hMN14 to Treat Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hMN14-03
Record Dates: First submitted 2002-07-11; First posted 2002-07-15 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2004-01

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Cancer; Pancreatic Carcinoma; Pancreatic Neoplasms; Pancreas Cancer; Pancreatic Tumor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — labetuzumab

INTERVENTIONS:
Drug: hMN14 (labetuzumab)

SUMMARY:
The purpose of this trial is to determine the safety of 90Y-hMN14 at different dose levels in the treatment of pancreatic cancer.

ELIGIBILITY:
Disease Characteristics:

* Patients with a documented histologic or cytologic diagnosis of a pancreatic malignancy
* Patients with recurrent, advanced and/or metastatic disease, who have either failed standard therapy or are not eligible for any alternate therapies of higher therapeutic priority.
* Patients with at least one identified (confirmed) and measureable tumor site.

Prior/Concurrent Therapy:

* Surgery: Patients are excluded if they have had major surgery either during or within four weeks prior to study entry.
* Chemotherapy: Patients must have failed standard therapy or are not eligible for any alternate therapies of higher therapeutic priority.
* Biologic Therapy: Patients who have received a chimeric, CDR-grafted (humanized), or human IgG will be eligible provided pre-study evaluations demonstrate no significant reactivity with hMN14 IgG (i.e., HAHA)
* Radiotherapy: No prior radiotherapy within four weeks of study entry. No prior external beam irradiation to a field that includes more than 30% of the red marrow. No prior radiation to maximal tolerable levels for any critical organ (e.g., 3,000 cGy for the liver; 2,000 cGy for the lungs and kidneys).
* Other: Any experimental therapy (i.e., drugs, biologics, procedures) for the primary malignancy, either during or within four weeks prior to study entry.

Patient Characteristics/Inclusion Criteria:

* Performance Status: Patients with a Karnofsky performance status > 70% (or equivalent, ECOG 0-1) and an expected survival rate of at least 3 months
* Hematopoietic: Hemoglobin > 10g/dL; WBC > 3000 per mm3; Granulocyte count > 1500 per mm3; platelet count > 100,000 per mm3
* Hepatic: Total bilirubin < 1.5 times the institutional upper limit of normal (IULN); AST or ALT < 2 X IULN
* Renal: Creatinine < IULN
* Cardiovascular: Patients with LVEF >/= 50% by required MUGA/2D-ECHO study
* Pulmonary: Patients with DF and FEV1 >/= 60 % by required Pulmonary Function Tests
* Gastrointestinal:Patients with severe anorexia or other related symptomology are excluded
* Central Nervous System: Patient with known metastatic disease to the CNS are excluded
* Other: Patients who have had a prior imaging study with a murine antibody may be included. Patients agreeing to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be preformed on each premenopausal female of childbearing potential immediately prior to entry into the study. Patients able to understand and give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2000-01; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, Study Chair — Gilead Sciences
Locations (10):
- United States (5):
  - Hoag Cancer Center, Newport Beach, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Bay Pines VA Medical Center, St. Petersburg, Florida
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
- Germany (2):
  - Medizinische Fakultaet der Charité Berlin, Berlin
  - Universitaetsklinikum Leipzig, Leipzig
- Hungary (2):
  - Semmelweis University, Budapest
  - Medical University of Szeged, Szeged
- Academic Medical Center, Amsterdam, Netherlands